CLINICAL TRIAL: NCT04265066
Title: Prehospital Analysis of the Sublingual Microvascular Terminal Circuit in Emergency Patients - a Prospective Observational Study
Brief Title: Microcirculation in Prehospital Medicine
Acronym: MicroCircPreHo
Status: Completed | Type: Observational
Sponsor: Klinik für Kardiologie, Pneumologie und Angiologie (Other)
Responsible Party: Sponsor-Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Principle Investigator Prof. Dr. Dr. Christian Jung, Heinrich-Heine University, Duesseldorf
Organization: Heinrich-Heine University, Duesseldorf (Other)
Other Study IDs: 16-031
Record Dates: First submitted 2020-01-29; First posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Emergencies
Keywords: Microcirculation; prehospital care; risk stratification
MeSH Terms: conditions — Emergencies | interventions — Microcirculation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Measurement of sublingual microcirculation
  Interventions: Diagnostic Test: microcirculation

INTERVENTIONS:
Diagnostic Test: microcirculation — measurement of microcirculation

SUMMARY:
Diagnostic and risk stratification are limited in emergencies. The measurement of microcirculation might identify patients with poor perfusion but compensated macrocirculation such as in beginning shock. This proof-of-concept study will examine whether sublingual prehospital sidestream dark field microscopy is feasible. This prospective observational study will include patients receiving medical aid by an emergency ambulance who had a spontaneous circulation and offer access to the sublingual mucosa. Sublingual measurement of microcirculation will be performed using a sidestream dark field camera. Video-quality will be evaluated with MIQS (microcirculation image quality score). AVA 4.3C software will calculate microcirculatory parameters.

DETAILED DESCRIPTION:
Risk stratification is a key element in emergency medicine and there is great interest to identify and validate novel tools and parameters. These tools must be are easy to handle even in the emergency setting by emergency physicians and paramedics. The main challenge for these tools is to identify critically ill patients, but usually, an ambulance disposes on clinical examination and basic hemodynamic values. Therefore, diagnostic tools are limited to the assessment of macrocirculatory values, which are not very reliable and might not necessarily reflect factual organ perfusion. Focusing only on macrocirculation might mask already ongoing impaired organ perfusion as tissue hypoxia is crucial and microcirculatory collapse or at least dysregulation occurs very early. Reduced microcirculation might result in attenuated cellular nutrient and oxygen supply that might result in severe cell damage. In fact, impaired microcirculation is ubiquitous in shock and can be found even in the setting of hemodynamic compensation. An impaired microcirculation is often the very first sign of alarm for deteriorating critically ill patients. A promising way to identify patients with impaired microcirculation is the use of sublingual IDF- and SDF-measurement (IDF: incident dark-field; SDF: sidestream dark field) devices as sublingual microcirculation is a suitable target because it reliably reflects organ perfusion. Measuring sublingual microcirculation has already been used to identify high-risk patients in many intra-hospital or experimental settings. These measurement tools are easy to use hand-held devices. The newest generation of SDF offers the great improvement of automatic software which independently calculates various microcirculatory parameters. Therefore, there is no need for the treating physician to interpret the videos by himself. This investigation will take place in the ambulance emergency service of the metropolitan area around Düsseldorf, Germany. To participate in the study, patients must meet the following criteria: 1) the call for an acute emergency outside the hospital with the indication for sending out an emergency doctor, 2) a spontaneous circulation without previous resuscitation, 3) informed consent, 4) the sublingual mucosa must be accessible. The following data will be collected: age, sex, cause for emergency alarm (cardiac reason, respiratory reason, gastroenterological, oncological, general internal medicine, renal, neurological, psychiatric, paediatric, traumatic), and the National Advisory Committee on Aeronautics' (NACA), that ranges from 0 = no injury, 7 = lethal injury severity score. Vital parameters (heart rate, non-invasive blood pressure, peripheral oxygen saturation) will be measured using a standard out-of-hospital monitoring device (Corpuls3 (GS Elektromedizinische Geräte G. Stemple GmbH, Kaufering, Germany)). Mean arterial pressure (MAP) will be calculated as follows: (2 * diastolic pressure + systolic pressure) /3. The capillary refill was evaluated in a standardized manner as described by Hernandez et al. Only sufficiently trained investigators will perform measurements. The microcirculation will be assessed by the implementation of the sidestream darkfield microscope (MicroScan® device, Microvision Medical, Amsterdam, The Netherlands). At the tip of the device, a highly sensitive camera digitally records the sublingual capillary network. The software analysis can directly be performed and visualized on a tablet screen. Additionally, the videos will be saved for later analysis. A suitable tablet computer will be used (Microsoft Surface Pro 4, (Redmond, Washington, USA). After acquisition of the videos, a validated automatic algorithm-software (AVA, Version 4.3 C) will perform the analyses. According to the second consensus on the assessment of sublingual microcirculation in critically ill patients (European Society of Intensive Care Medicine), the following parameters of microcirculation will be assessed both for all and for small vessels: PPV (Percentage of Perfused Vessels), NC (Number of Crossings), PNC (Perfused Number of crossings), TVD (Total Vessel Density), PVD (Perfused Vessel Density). The study plans to include at least 25 patients.

ELIGIBILITY:
Inclusion Criteria:

* the call for an acute emergency outside the hospital with the indication for sending out an emergency doctor
* a spontaneous circulation without previous resuscitation
* informed consent
* the sublingual mucosa must be accessible

Exclusion Criteria:

* <18 years
* Lacking informed consent
* time-critical disease
* previous resuscitation
* inaccessibility of sublingual area

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who call for an acute emergency outside the hospital
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Microcirculatory quality score (MIQS) | at Baseline
  MIQS by Massey et al. is an established method to validate recorded SDF-videos for their suitability for further analysis. MIQS assigns a score of optimal (0 points), suboptimal but acceptable (1 point), or unacceptable (10 points) to the categories illumination, duration, focus, content, stability, and pressure. The scoring will be done for every recorded video during the offline analysis.
Percentage of Perfusion Vessels [%] | at Baseline
  Measurement of sublingual microcirculation by using MicroScan® microscope. AVA 4.3C calculates automatically important microcirculatory values (Percentage of Perfusion Vessels; DeBackerDensity; Perfused DeBackerDensity; Perfused Vessel Density) according to the Second Consensus Conference

SECONDARY OUTCOMES:
NACA-scores | at Baseline
  The National Advisory Committee on Aeronautics' (NACA) score ranges from 0 = no injury, 7 = lethal injury severity score and is an established method to estimate the severity of disease of emergency patients.
measurement of Blood pressure | at Baseline
  Non-invasive blood-measurement will be done immediately for every emergency patient.
measurement of Pulse rate [/per Minute] | at Baseline
  Non-invasive pulse rate-measurement will be done immediately for every emergency patient using a pulsoxymeter.
measurement of Peripheral oxygen saturation [%] | at Baseline
  Non-invasive oxygen saturation measurement will be done immediately for every emergency patient using a pulsoxymeter.
measurement of Respiratory rate [/Minute] | at Baseline
  Respiratory rate will be assessed visually for every emergency patient
measurement of microcirculation | at Baseline
  Measurement of sublingual microcirculation by using MicroScan® microscope
Intra-Hospital Mortality | up to 1 year
  Intra-Hospital mortality will be assessed using the medical records of the hospital or direct contact to the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Pulmonary Disease and Vascular Medicine, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: Undecided